CLINICAL TRIAL: NCT05495893
Title: Mycophenolate Mofetil Versus Cyclophosphamide in the Induction Therapy of Pediatric Patients With Active Proliferative Lupus Nephritis: A Prospective, Randomized, Multicenter, Open-label, Parallel-arm Study
Brief Title: MMF Versus CYC in the Induction Therapy of Pediatric Active Proliferative LN
Acronym: MyCITS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Beijing Children's Hospital (Other); Jiangxi Province Children's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Shenzhen Children's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Xiaochuan Wu, Director of Pediatrics, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021YFC2702004
Record Dates: First submitted 2022-07-25; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Mycophenolate Mofetil; Cyclophosphamide; Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide (Experimental): Cyclophosphamide for injection, 750mg/m2 each time, 1g at most, once a month for 6 consecutive months. Steroids : intravenous methylprednisolone, 15~30mg/kg · day, maximum 1000mg/day, 3 consecutive days a week for 2 weeks; during the interval of methylprednisolone pulse therapy and after:prednisone tablets 2mg/kg · day with a maximum dose 60mg / day
  Interventions: Drug: Cyclophosphamide
- Mycophenolate mofetil (Experimental): Mycophenolate mofetil, tablets, 30-40mg/ (kg · day), BID, the maximum amount is no more than 2g/d. Steroids : intravenous methylprednisolone, 15~30mg/kg · day, maximum 1000mg/day, 3 consecutive days a week for 2 weeks; during the interval of methylprednisolone pulse therapy and after:prednisone tablets 2mg/kg · day with a maximum dose 60mg / day
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Cyclophosphamide — The patients will be divided into two groups randomly. Cyclophosphamide for injection, 750mg/m2 each time, 1g at most, once a month for 6 consecutive months. Steroids : intravenous methylprednisolone, 15~30mg/kg · day, maximum 1000mg/day, 3 consecutive days a week for 2 weeks; during the interval of methylprednisolone pulse therapy and after:prednisone tablets 2mg/kg · day with a maximum dose 60mg / day. The duration of induction therapy: 6 months.
  Arms: Cyclophosphamide
Drug: Mycophenolate Mofetil — The patients will be divided into two groups randomly. Mycophenolate mofetil, tablets, 30-40mg/ (kg · day), BID, the maximum amount is no more than 2g/d. Steroids : intravenous methylprednisolone, 15~30mg/kg · day, maximum 1000mg/day, 3 consecutive days a week for 2 weeks; during the interval of methylprednisolone pulse therapy and after:prednisone tablets 2mg/kg · day with a maximum dose 60mg / day. The duration of induction therapy: 6 months.
  Arms: Mycophenolate mofetil

SUMMARY:
A prospective, randomized, multicenter, open-label, parallel-arm Study to compare effectiveness of mycophenolate mofetil versus cyclophosphamide in the Induction Therapy of pediatric patients with Active Proliferative Lupus Nephritis in Chinese population

DETAILED DESCRIPTION:
Scattered research in adults showed that both mycophenolate mofetil (MMF) and cyclophosphamide (CYC) can be used in the induction therapy of lupus nephritis. however data is limited in children.Therefore, the purpose of this study is to observe and compare the efficacy and safety of MMF and CYC as induction therapy for children with proliferative lupus nephritis through a multi-center open randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

Only those who fully meet the following criteria can be considered for inclusion in this study:

1. Age 5-17 years old;
2. SLE patients who meet the updated 2019 eular/acr SLE classification criteria or 2012 SLICC diagnostic criteria;
3. According to the revised International Society of Nephrology / Society of renal pathology (isn/rps) classification in 2018, it conforms to active proliferative ln type III or IV, with or without type V;
4. Glomerular filtration rate EGFR ≥ 60 ml/min/1.73 m2;
5. 24-hour urinary protein quantitation ≥ 25mg/kg, or urinary protein / creatinine 1.0mg/mg;
6. Blood routine WBC count ≥ 3.0*10^9/l, lymphocyte ≥ 0.5*10^9/l before enrollment;
7. No immunosuppressants such as cyclophosphamide, mycophenolate mofetil, cyclosporine A, tacrolimus, azathioprine, methotrexate, or biological agents such as rituximab, baileyoumab, and etaxel were used before enrollment.

Exclusion Criteria:

1. A known history of primary immunodeficiency, splenectomy, or any potential disease that makes participants vulnerable to infection;
2. Evidence of hepatitis C, active hepatitis B, HIV infection, tuberculosis infection, severe fungal infection, or other serious infections;
3. Have any history of tumor or cancer;
4. Patients with lupus encephalopathy, diffuse alveolar hemorrhage, severe hemolytic anemia, blood routine platelet count lower than 10.0*10^9/l, glomerular filtration rate eGFR < 60 ml/min/1.73 m2, or patients with other serious complications have unstable vital signs;
5. Have severe gastrointestinal bleeding, pancreatitis, serious heart, liver, blood, endocrine system diseases;
6. Patients who are known to be allergic to mycophenolate mofetil, cyclophosphamide, glucocorticoids or any of the above drugs;
7. Patients who participated in other clinical trials within 3 months before enrollment;
8. The researcher judged that the patient's condition was not suitable for participants in this trial.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Effective rate of LN treatment | 6 months
  complete remission and partial remission

SECONDARY OUTCOMES:
complete remission time | 6 months
  complete remission time within 6 months of designed induction therapy
Incidence of LN treatment failure | 6 months
  occurrence of end stage renal disease or serum creatinine reached twice the baseline or 24 urinary protein or urinary protein / creatinine reached twice the baseline at 6 months of follow-up.
Incidence of creatinine doubling | 6 months
  serum creatinine reaching 2 times of the baseline level
LN recurrence rate | 6 months
  (1) proteinuria recurrence, which is defined as continuous proteinuria ≥ 1.0 g/d (or 25mg/kg) after complete remission (CR) or increase ≥ 2.0 g/d (or 50mg/d) after partial remission (PR), with or without hematuria; (2) The increase of Scr level is defined as the increase of Scr level ≥ 50% when the baseline examination is normal, or 30% when the baseline examination is abnormal.
SLE recurrence rate | 6 months
  new onset of skin erythema, vasculitis, joint pain, hematological diseases (platelet <50*109/l or hemolytic anemia), neurological symptoms, lupus myocarditis, lupus pneumonia, serous cavity inflammation or new abnormalities in laboratory examination (antibodies, C3 and C4), and SLEDAI score greater than or equal to 4 points.
SLE disease activity score | 6 months
  Systemic Lupus Erythematosus Disease Activity Index 2000 score at 6 months
partial remission time | 6 months
  Partial remission time within 6 months of designed

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochuan Wu, Study Chair — The Second Xiangya Hospital, Central South University
Locations (1):
- the Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No